CLINICAL TRIAL: NCT00620490
Title: Postoperative Analgesia After Thoracotomy Without Thoracic Epidural Analgesia : Paravertebral Analgesia With a Catheter Associated With Intravenous Morphine Patient-controlled-analgesia (Pca)
Brief Title: Paravertebral Analgesia Associated With Intravenous Morphine PCA After Thoracotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4068
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Pain
Keywords: Epidural analgesia; Contraindications; Paravertebral nerve block analgesia; ropivacaine; Visual analogical scale; Morphine; Side effects; Pain and thoracotomy
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ropivacaine 0.5% 0.1 ml/kg per hour
  Interventions: Drug: ropivacaine
- 2 (Placebo Comparator)
  Interventions: Other: nacl 0,9%

INTERVENTIONS:
Drug: ropivacaine — Ropivacaine 0.5% 0.1 ml/kg per hour
  Arms: 1
Other: nacl 0,9% — saline 0.9% 0.1 ml/kg per hour
  Arms: 2

SUMMARY:
osteolateral thoracotomy is a painful surgical procedure.Thoracic epidural analgesia (TEA) is usually considered as the "gold standard" for postoperative thoracic analgesia. Unfortunately, it's not always possible to realize it because of contraindications or because of technical failures.Analgesia using a paravertebral block is an alternative to the TEA : it provides an unilateral sensitive and sympathetic block using a catheter.In our study, the catheter will be placed by the thoracic surgeon at the end of the surgical procedure, under direct vision, to insure maximal security also on patients on antiplatelets agents, anticoagulants or with haemostasis disorders (the placement of the catheter by the anaesthetist with the loss of resistance technique is contraindicated in these cases).Patients will be randomized to receive either a continuous 48-hours infusion of ropivacaine 0,5% or saline serum in the control group.All patients are connected to a PCA pump with intravenous morphine and will receive paracetamol and nefopam.The visual analogic scale (VAS) at rest and on movement, total morphine consumption and side effects will be recorded during the first 48 hours after surgery. The aim of this study is to prove a decrease of pain at rest and on movement, a decrease of the cumulated total morphine dose consumption and a decrease of the side effects (nausea, vomiting, pruritus, sedation, bradypnea, urinary retention).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracotomy who presented with contraindications to TEA.Contraindications to TEA are :
* Patient's refusal after informations about advantages and risks of the technique
* Anti platelets treatment that can't be discontinued
* Anticoagulants at a curative dosage- haemostasis and/or coagulation disorders: thrombopenia < 100.000/mm3, ACT > 1,5 / control, PTT < 75%- Systemic or local infection of the puncture point
* 2 and 3 grade atrio-ventricular heart block without pacing
* Severe aortic valve stenosis
* Kyphoscoliosis
* certain neurological disorders

Exclusion Criteria:

* Patient's refusal to participate in the study
* Psychiatric disorder (impossibility to collect the informed consent)
* Patient under juridical protection
* On going an other study
* Pregnancy, breastfeeding
* Non balanced epilepsy
* 3 grade auriculae-ventricular heart block without pacing
* Severe hepatocellular insufficiency
* Anti arrhythmic treatment : class III of the Vaughan William's classification- Skin infection of the puncture point
* Allergy to aminoamides local anaesthetic
* Surgical difficulties to insert paravertebral catheter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain after surgery | first 48 hours after surgery

SECONDARY OUTCOMES:
· Total dosis of morphine consumption, side effects nausea, vomiting,pruritus,Urinary retention, respiratory rate and sedation, · heart rate, blood pressure and peripheral saturation | first 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Helms, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Chirurgie Thoracique, Hôpitaux Universitaires, Strasbourg, France

REFERENCES:
- [Result] Helms O, Mariano J, Hentz JG, Santelmo N, Falcoz PE, Massard G, Steib A. Intra-operative paravertebral block for postoperative analgesia in thoracotomy patients: a randomized, double-blind, placebo-controlled study. Eur J Cardiothorac Surg. 2011 Oct;40(4):902-6. doi: 10.1016/j.ejcts.2011.01.067. Epub 2011 Mar 5. PMID 21377888